CLINICAL TRIAL: NCT04849299
Title: A Phase 1, Randomized, Open-Label Study to Evaluate the Effect of Cyclosporine on the Plasma Pharmacokinetics of AT-527 in Healthy Adult Male Subjects
Brief Title: Effect of Cyclosporine on the Pharmacokinetics (PK) of AT-527 (R07496998)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-005
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT-527 550 mg + cyclosporine (simultaneous) (Experimental): n=12
  Interventions: Drug: AT-527 550 mg + cyclosporine
- AT-527 550 mg + cyclosporine (staggered) (Experimental): n=12
  Interventions: Drug: AT-527 550 mg + cyclosporine

INTERVENTIONS:
Drug: AT-527 550 mg + cyclosporine — 550 mg AT-527 alone on Day 1 and 550 mg AT-527 plus 600 mg cyclosporine administered simultaneously on Day 7 Other Names: AT-527 is also known as R07496998
  Arms: AT-527 550 mg + cyclosporine (simultaneous)
Drug: AT-527 550 mg + cyclosporine — 550 mg AT-527 alone on Day 1 and 550 mg AT-527 plus 600 mg cyclosporine administered on Day 7 (with dosing offset by 2 hrs) Other Names: AT-527 is also known as R07496998
  Arms: AT-527 550 mg + cyclosporine (staggered)

SUMMARY:
This study will determine the effect of cyclosporine on the PK of AT-527 (R07496998) in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Concomitant use of prescription medications, or systemic over-the-counter medications
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy adult male subjects
Enrollment: 24 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 (R07496998): Cmax | Day 1 vs Day 7
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of AT-527 (R07496998): AUC | Day 1 vs Day 7
  Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Montreal, Quebec, Canada